CLINICAL TRIAL: NCT03822468
Title: A Phase II, Multicenter, Randomized, Open-label Study to Evaluate the Safety and Efficacy of 400 mg of Ribociclib in Combination With Non-steroidal Aromatase Inhibitors for the Treatment of Pre- and Postmenopausal Women With Hormone Receptor-positive, HER2-negative Advanced Breast Cancer Who Received no Prior Therapy for Advanced Disease
Brief Title: Study of 2 Ribociclib Doses in Combination With Aromatase Inhibitors in Women With HR+, HER2- Advanced Breast Cancer
Acronym: AMALEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011A2207; 2018-004234-15 (EudraCT Number)
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer (BC); hormone receptor (HR); HR-positive; human epidermal growth factor receptor 2 (HER2); HER2-negative; ER-positive; advanced breast cancer (aBC); ribociclib (LEE011); premenopausal; postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Anastrozole; Letrozole; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib 400 mg (Experimental): Ribociclib 400 mg QD 3 weeks on/1 week off + letrozole or anastrozole (+goserelin in premenopausal women)
  Interventions: Drug: Ribociclib; Drug: Anastrozole; Drug: Letrozole; Drug: Goserelin
- Ribociclib 600 mg (Active Comparator): Ribociclib 600 mg QD 3 weeks on/1 week off + letrozole or anastrozole (+ goserelin in premenopausal women)
  Interventions: Drug: Ribociclib; Drug: Anastrozole; Drug: Letrozole; Drug: Goserelin

INTERVENTIONS:
Drug: Ribociclib — Ribociclib (at a dosage of 400 mg or 600 mg) QD orally taken on days 1 to 21 of a 28-day cycle, followed by 7 days off ribociclib (days 22 to 28). Ribociclib was supplied as 200 mg tablets as individual patient supply packaged bottles.
  Other Names: LEE011
Drug: Anastrozole — Anastrozole 1 mg tablets for oral use QD continuously
Drug: Letrozole — Letrozole 2.5 mg tablets for oral use QD continuously
Drug: Goserelin — Goserelin 3.6 mg subcutaneously once every 4 weeks (pre-menopausal women only)

SUMMARY:
The purpose of the study was to evaluate the safety and efficacy of a reduced ribociclib starting dose of 400 mg in combination with a non-steroidal aromatase inhibitor (NSAI) (letrozole or anastrozole) for the treatment of pre- and postmenopausal women with hormone receptor-positive (HR-positive), HER2-negative advanced breast cancer (aBC) who have received no prior therapy for advanced disease. Premenopausal women were required to receive goserelin in both treatment arms.

DETAILED DESCRIPTION:
Patients were assigned at visit Cycle 1 Day 1 to one of the following two treatment arms in a ratio of 1:1:

* Experimental arm: Ribociclib 400 mg (2 × 200 mg tablets by mouth) QD on Days 1 to 21 of a 28-day cycle, followed by 7 days off ribociclib (Days 22 to 28) in combination with ET consisting of:

  • For postmenopausal women:
  * Letrozole 2.5 mg by mouth QD continuously or anastrozole 1 mg by mouth QD continuously

    • For premenopausal women:
  * Letrozole 2.5 mg by mouth QD continuously or anastrozole 1 mg by mouth QD continuously, combined with goserelin 3.6 mg subcutaneously once every 4 weeks.
* Control arm: Ribociclib 600 mg (3 × 200 mg tablets by mouth) QD on Days 1 to 21 of a 28-day cycle, followed by 7 days off ribociclib (Days 22 to 28) in combination with ET consisting of:

  * For postmenopausal women:

    ~ Letrozole 2.5 mg by mouth QD continuously or anastrozole 1 mg by mouth QD continuously.
  * For premenopausal women:

    * Letrozole 2.5 mg by mouth QD continuously or anastrozole 1 mg by mouth QD continuously, combined with goserelin 3.6 mg subcutaneously once every 4 weeks.

Participants received study treatment until disease progression (radiologically documented according to RECIST 1.1 criteria), unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

For participants who discontinued treatment for reasons other than documented disease progression, death, lost to follow-up, or withdrawal of consent, tumor assessments continued to be performed until disease progression, death, lost to follow-up, or withdrawal of consent (post-treatment efficacy follow-up).

ELIGIBILITY:
Key inclusion criteria:

* Patient has advanced (loco-regionally recurrent or metastatic) breast cancer not amenable to curative therapy.
* Patient has a histologically and/or cytologically confirmed diagnosis of ER-positive and/or PgR-positive breast cancer based on the most recently analyzed tissue sample, and all tested by local laboratory.
* Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing and based on the most recently analyzed tissue sample.
* Patient must have measurable disease, i.e., at least one measurable lesion according to RECIST version 1.1. (a lesion in a previously irradiated site may only be counted as a target lesion if there is clear evidence of progression since the irradiation).
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Standard 12-lead ECG values defined as the mean of the triplicate ECGs and assessed by the central laboratory:

  * QTcF interval at screening < 450 ms (QT interval using Fridericia's correction)
  * Mean resting heart rate 50 to 90 bpm (determined from the ECG)
* Women of childbearing potential (CBP), defined as all women physiologically capable of becoming pregnant, must have confirmed negative serum pregnancy test (for β-hCG) within 14 days prior to randomization.
* Women of CBP must be willing to use highly effective methods of contraception.

Key Exclusion Criteria:

* Patient with symptomatic visceral disease or any disease burden that makes the patient ineligible for endocrine therapy per the investigator's judgment.
* Patient who received any prior systemic anti-cancer therapy(including endocrine therapy, chemotherapy, prior CDK4/6 inhibitors) for aBC. Patients who received neo-/adjuvant therapy for breast cancer are eligible.
* Patient is concurrently using other anti-cancer therapy.
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major toxicities.
* Patient has received extended-field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to randomization, and has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion). Patients in whom ≥
* 25% of the bone marrow has been previously irradiated are also excluded.
* Patient has a concurrent malignancy or malignancy within 3 years of the randomization date, with the exception of adequately treated basal or squamous cell skin carcinoma, or curatively resected cervical carcinoma in situ.
* Patients with central nervous system (CNS) involvement unless they meet specific stability criteria.
* Patient has clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality.
* Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, and has not fully recovered from side effects of such treatment.

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (83):
- United States (14):
  - Southern Cancer Center PC, Mobile, Alabama
  - Marin Cancer Care, Greenbrae, California
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Florida Retina Institute, Orlando, Florida
  - Weinberg Cancer Institute at FSH, Baltimore, Maryland
  - Nebraska Hematology Oncology P C, Lincoln, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Cntr Of Nevada, Henderson, Nevada
  - New York Oncology Hematology, Albany, New York
  - Mount Sinai School Of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Millennium Research Clin Develop, Houston, Texas
  - Texas Oncology, McAllen, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Novartis Investigative Site, San Juan, Argentina
- Austria (4):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Namur
- Brazil (5):
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Goiânia
  - Novartis Investigative Site, São José do Rio Preto
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Novartis Investigative Site, Cambridge, Ontario, Canada
- Colombia (4):
  - Novartis Investigative Site, Valledupar, Cesar Department
  - Novartis Investigative Site, Ibagué, Tolima Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Montería
- Novartis Investigative Site, San José, Costa Rica
- Czechia (2):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Prague
- Finland (2):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
- France (9):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lyon 08
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Valenciennes
- Germany (8):
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Weiden
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szolnok
- India (5):
  - Novartis Investigative Site, Raipur, Chhattisgarh
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Bhubaneshwar, Odisha
  - Novartis Investigative Site, Delhii
  - Novartis Investigative Site, Mumbai
- Novartis Investigative Site, Amman, Jordan
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Peru (4):
  - Novartis Investigative Site, Trujillo, La Libertad
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
- Portugal (3):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Loures
  - Novartis Investigative Site, Porto
- Russia (3):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Parktown
- Sweden (2):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Cardoso F, Jacot W, Kuemmel S, Gupta S, Cruz F, Balaraman R, Ferreira A, Ahola T, Chapko Y, Zhukova L, Chiang W, Li Z, Ji Y, Kaakiou N, Bolotova N, Sparano JA. 600- vs 400-mg First-Line Ribociclib in Hormone Receptor-Positive/ERBB2-Negative Advanced Breast Cancer: The AMALEE Randomized Clinical Trial. JAMA Oncol. 2025 Nov 1;11(11):1356-1363. doi: 10.1001/jamaoncol.2025.3687. PMID 40996770
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 90 centers across 23 countries.
Pre-assignment Details: A total of 558 subjects were screened of which 376 participants were randomized on a 1:1 basis.
Period: Treatment Period
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Started | 188 | 188
Completed | 0 | 0
Not Completed | 188 | 188
Not completed — Progressive disease | 98 | 94
Not completed — Adverse Event | 21 | 24
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Physician Decision | 9 | 7
Not completed — Protocol Violation | 2 | 1
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Sponsor decision | 46 | 53
Period: Post-treatment Efficacy Follow-up
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Started | 22 | 26
Completed | 0 | 0
Not Completed | 22 | 26
Not completed — Progressive disease | 11 | 14
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Sponsor decision | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg | Total
Number analyzed (Participants) | 188 | 188 | 376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (12.96) | 57.0 (12.37) | 57.9 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 188 | 376
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 147 | 143 | 290
  Native American or Alaska Native | 14 | 10 | 24
  Asian | 13 | 9 | 22
  Black | 5 | 12 | 17
  Other | 1 | 4 | 5
  Unknown | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR defined as the percentage of participants with best overall response (BOR) of confirmed complete response (CR) or partial response (PR) assessed by local investigators according to RECIST 1.1.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 23.8 months
Population: The Full Analysis Set (FAS) including all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 188 | 188
Percentage of participants | 41.5 [34.4 to 48.7] | 45.3 [38.1 to 52.6]

2. Secondary Outcome: Change From Baseline in QTc (With Fridericia's Correction) at Cycle 1 Day 15 (at 2 Hours Post-dose)
Description: Electrocardiogram (ECG) data was collected via 12-lead digital ECG machines. Change from baseline in the QT interval (a segment of the ECG that reflects the time it takes for the heart to repolarize after each heartbeat) was corrected for heart rate using Fridericia's formula (ΔQTcF).
Time Frame: Baseline and Cycle 1 Day 15 at 2 hours post-dose. Cycle = 28 days
Population: Participants who received at least one dose of study treatment and had available QT assessments conducted at both baseline and Cycle 1 Day 15 (2 hours post-dose)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 174 | 175
milliseconds | 12.5 (12.91) | 19.7 (18.50)

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) was defined as the time from the date of randomization to the date of the first documented disease progression or death due to any cause. PFS was censored if no PFS event was observed. The censoring date was the date of the last adequate tumor assessment. Clinical deterioration without objective radiological evidence was not considered as documented disease progression. PFS was assessed via a local radiology assessment as well as Blinded Independent Review Committee (BIRC) according to RECIST 1.1.
Time Frame: Up to approximately 60 months
Population: The Full Analysis Set (FAS) including all randomized participants
Measure: Median (Full Range); unit: Months
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 188 | 188
Months | 26.9 [20.3 to 30.4] | 25.1 [19.4 to 33.4]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) was defined as the proportion of patients with a best overall response of complete response (CR), or partial response (PR), or an overall response of stable disease (SD), lasting for at least 24 weeks. CR, PR, and SD were defined as per local review as well as Blinded Independent Review Committee (BIRC) according to RECIST 1.1. A patient was considered to have SD for 24 weeks or longer if a SD response was recorded at 24-1=23 weeks or later from randomization, allowing for the ±1 week visit window for tumor assessments.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 60 months
Population: The Full Analysis Set (FAS) including all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 188 | 188
Participants | 142 | 133

5. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) was defined as the time from the date of randomization to the first documented response of either complete response (CR) or partial response (PR), which had to be subsequently confirmed (although the date of initial response was used, not the date of confirmation). CR and PR were based on tumor response data as per local review and according to RECIST 1.1.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 60 months
Population: Full Analysis Set (FAS) - Only responders included
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 90 | 103
Months | 13.1 [7.4 to NA] — NA: Not estimable due to insufficient number of participants with events | 9.0 [5.6 to 16.4]

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) only applied to patients whose best overall response was complete response (CR) or partial response (PR) according to RECIST 1.1 based on tumor response data per local review. The start date was the date of first documented response of CR or PR (i.e. the start date of response, not the date when response was confirmed), and the end date was defined as the date of the first documented progression or death due to underlying cancer. Patients continuing without progression or death due to underlying cancer were censored at the date of their last adequate tumor assessment.
  CR: Disappearance of all lesions with lymph nodes measuring < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 60 months
Population: Full Analysis Set (FAS) - Only responders included
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 90 | 103
Months | 26.5 [16.8 to NA] — NA: Not estimable due to insufficient number of participants with events | 28.8 [22.6 to NA] — NA: Not estimable due to insufficient number of participants with events

7. Secondary Outcome: Pharmacokinetics (PK) of Ribociclib: Maximum Observed Plasma Concentration (Cmax)
Description: PK parameters were calculated by non-compartmental analysis. Cmax is the maximum observed plasma drug concentration after single dose administration.
Time Frame: Cycle 1 Day 15 at pre-dose, and 2, 4, 6 and 24 hours post-dose. Cycle = 28 days
Population: Participants who provided an evaluable PK parameter (Cmax) and received at least 10 consecutive daily ribociclib doses of 400 mg or 600 mg immediately prior to and on the PK collection day
Measure: Mean (Standard Deviation); unit: nanogram / milliliter (ng / mL)
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 20 | 16
nanogram / milliliter (ng / mL) | 1240 (739) | 1740 (918)

8. Secondary Outcome: PK of Ribociclib: Time to Reach Observed Maximum Concentration (Tmax)
Description: PK parameters were calculated by non-compartmental analysis. Tmax is the time to reach maximum observed plasma concentration. Actual recorded sampling times were considered for the calculations.
Time Frame: Cycle 1 Day 15 at pre-dose, and 2, 4, 6 and 24 hours post-dose. Cycle = 28 days
Population: Participants who provided an evaluable PK parameter (Tmax) and received at least 10 consecutive daily ribociclib doses of 400 mg or 600 mg immediately prior to and on the PK collection day
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 20 | 16
hours (h) | 2.08 [1.83 to 4.38] | 4.00 [1.83 to 23.8]

9. Secondary Outcome: PK of Ribociclib: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC0-24)
Description: PK parameters were calculated by non-compartmental analysis. AUC0-24 is the area under the plasma concentration-time curve from 0 to 24 hours
Time Frame: Cycle 1 Day 15 at pre-dose, and 2, 4, 6 and 24 hours post-dose. Cycle = 28 days
Population: Participants who provided an evaluable PK parameter (AUC0-24) and received at least 10 consecutive daily ribociclib doses of 400 mg or 600 mg immediately prior to and on the PK collection day
Measure: Mean (Standard Deviation); unit: ng x h / mL
Arm/Group | Ribociclib 400 mg | Ribociclib 600 mg
Number analyzed (Participants) | 17 | 13
ng x h / mL | 18700 (11600) | 31600 (14300)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first dose of study treatment to 30 days after last dose of study medication (on-treatment), up to 23.8 months. Deaths were collected in the post-treatment efficacy follow-up from 31 days after last dose of study medication until the end of the study, up to 62 months.
Description: Deaths in the post-treatment efficacy follow-up were not considered adverse events. The total number at risk in the post-treatment efficacy follow-up included patients who entered this period.
Groups:
- Ribociclib 400mg: Ribociclib 400 mg QD 3 weeks on/1 week off + letrozole or anastrozole (+goserelin in premenopausal women) - Events up to 30 days safety follow-up
- Ribociclib 600mg: Ribociclib 600 mg QD 3 weeks on/1 week off + letrozole or anastrozole (+ goserelin in premenopausal women) - Events up to 30 days safety follow-up
- Ribociclib 400mg (Post-treatment Efficacy Follow-up): Ribociclib 400mg (Post-treatment efficacy follow-up) - Deaths in the post-treatment efficacy follow-up period were not considered adverse events.
- Ribociclib 600 mg (Post-treatment Efficacy Follow-up): Ribociclib 600 mg (Post-treatment efficacy follow-up) - Deaths in the post-treatment efficacy follow-up period were not considered adverse events.
Arm/Group | Ribociclib 400mg | Ribociclib 600mg | Ribociclib 400mg (Post-treatment Efficacy Follow-up) | Ribociclib 600 mg (Post-treatment Efficacy Follow-up)
All-Cause Mortality (participants affected / at risk) | 5/188 | 6/188 | 3/22 | 2/26
Serious Adverse Events (participants affected / at risk) | 38/188 | 37/188 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 175/188 | 178/188 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib 400mg (N=188) | Ribociclib 600mg (N=188) | Ribociclib 400mg (Post-treatment Efficacy Follow-up) (N=0) | Ribociclib 600 mg (Post-treatment Efficacy Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 2 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | NA | NA
Colitis (Gastrointestinal disorders) | 2 | 0 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | NA | NA
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Ileus (Gastrointestinal disorders) | 1 | 0 | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 1 | 1 | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 1 | NA | NA
Asthenia (General disorders) | 0 | 1 | NA | NA
Ill-defined disorder (General disorders) | 0 | 1 | NA | NA
Pain (General disorders) | 1 | 1 | NA | NA
Pyrexia (General disorders) | 1 | 0 | NA | NA
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 1 | NA | NA
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0 | NA | NA
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | NA | NA
COVID-19 (Infections and infestations) | 2 | 2 | NA | NA
COVID-19 pneumonia (Infections and infestations) | 3 | 1 | NA | NA
Cellulitis (Infections and infestations) | 1 | 0 | NA | NA
Coronavirus pneumonia (Infections and infestations) | 1 | 0 | NA | NA
Diverticulitis (Infections and infestations) | 1 | 1 | NA | NA
Lymphangitis (Infections and infestations) | 0 | 2 | NA | NA
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | NA | NA
Pneumonia (Infections and infestations) | 2 | 3 | NA | NA
Postoperative wound infection (Infections and infestations) | 1 | 0 | NA | NA
Sepsis (Infections and infestations) | 1 | 1 | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 0 | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Radiation injury (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Blood bilirubin increased (Investigations) | 1 | 0 | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | NA | NA
Hydrocephalus (Nervous system disorders) | 1 | 0 | NA | NA
Seizure (Nervous system disorders) | 1 | 0 | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | NA | NA
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | NA | NA
Depression (Psychiatric disorders) | 2 | 0 | NA | NA
Disorientation (Psychiatric disorders) | 0 | 1 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 1 | NA | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 1 | NA | NA
Embolism (Vascular disorders) | 1 | 0 | NA | NA
Peripheral embolism (Vascular disorders) | 1 | 0 | NA | NA
Venous thrombosis (Vascular disorders) | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib 400mg (N=188) | Ribociclib 600mg (N=188) | Ribociclib 400mg (Post-treatment Efficacy Follow-up) (N=0) | Ribociclib 600 mg (Post-treatment Efficacy Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 31 | 49 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 40 | 52 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 17 | 18 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 100 | 125 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 19 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 10 | 12 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 5 | 12 | NA | NA
Constipation (Gastrointestinal disorders) | 17 | 21 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 22 | 25 | NA | NA
Nausea (Gastrointestinal disorders) | 31 | 44 | NA | NA
Vomiting (Gastrointestinal disorders) | 15 | 22 | NA | NA
Asthenia (General disorders) | 24 | 23 | NA | NA
Fatigue (General disorders) | 22 | 40 | NA | NA
Oedema peripheral (General disorders) | 8 | 12 | NA | NA
Pain (General disorders) | 1 | 14 | NA | NA
Pyrexia (General disorders) | 11 | 12 | NA | NA
COVID-19 (Infections and infestations) | 17 | 27 | NA | NA
Nasopharyngitis (Infections and infestations) | 6 | 12 | NA | NA
Urinary tract infection (Infections and infestations) | 15 | 17 | NA | NA
Alanine aminotransferase increased (Investigations) | 49 | 47 | NA | NA
Aspartate aminotransferase increased (Investigations) | 41 | 40 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 11 | 17 | NA | NA
Blood creatinine increased (Investigations) | 12 | 15 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 14 | 26 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 17 | 16 | NA | NA
Lipase increased (Investigations) | 9 | 12 | NA | NA
Neutrophil count decreased (Investigations) | 25 | 24 | NA | NA
Weight decreased (Investigations) | 11 | 11 | NA | NA
White blood cell count decreased (Investigations) | 13 | 22 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 11 | 13 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 12 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 15 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 10 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 10 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 28 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 23 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 17 | NA | NA
Headache (Nervous system disorders) | 18 | 31 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 23 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 15 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 24 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 15 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 17 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 7 | 16 | NA | NA
Hot flush (Vascular disorders) | 24 | 14 | NA | NA
Hypertension (Vascular disorders) | 6 | 10 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03822468/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT03822468/SAP_001.pdf